CLINICAL TRIAL: NCT07261332
Title: A Comparative Study on Early Versus Delayed Induction of Labour in Patients With Prelabour Rupture of Membranes at Term
Brief Title: Early V/S Delayed Induction of Labour in Patients With Prelabour Rupture of Membranes
Acronym: PROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laiba Qamar (Other)
Responsible Party: Sponsor-Investigator, Laiba Qamar, Supervisor, University of Health Sciences Lahore
Organization: University of Health Sciences Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #PLROM225#
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Prelabor Rupture of Membranes; Labor (Obstetrics)--Complications; Induction of Labor
Keywords: prelabor rupture of membranes; complicated labor; early Versus delayed labor induction
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early induction of labour for PROM (Experimental): The patients assigned with this arm when presented with PROM were inducted immidiately for labour and no observation was done for 24 hours for spontaneous induction of labour
  Interventions: Drug: 0.5mg PGE2 gel
- Late induction of Labour in PROM (Active Comparator): The patients assigned with this arm were observed for 24 hours for any spontanous induction of labour and then only proceeded with manual induction.
  Interventions: Drug: 0.5mg PGE2 gel

INTERVENTIONS:
Drug: 0.5mg PGE2 gel — In this interventional group patients presenting with PROM will be immediately induced by 0.5mg PGE2 gel. If bishop score will not improve after 6 hours, then application of PGE2 gel will be repeated (maximum 2 doses)
  Arms: early induction of labour for PROM
Drug: 0.5mg PGE2 gel — The patients assigned with this intervention will be observed for 24 hours following which induction will be done using 0.5mg PGE2 gel in posterior fornix of vagina.
  Arms: Late induction of Labour in PROM

SUMMARY:
To compare the effects of early V/s delayed induction of labour and its outcomes in patients presenting with PROM without labour.

DETAILED DESCRIPTION:
This is a comparative study where the patient who presented with PROM were assigned 2 groups of intervention . One had early induction of labour and other had induction of labour after 24 hours of observation. Both groups were compared for the average time of labour till delivery of the fetus and the frequency of spontaneous vaginal delivery was also calculated for each group.

ELIGIBILITY:
Inclusion Criteria:

1. singleton pregnancy with cephalic presentation
2. gestational age between 37-41 weeks as calculated by last menstrual period date or early dating ultrasoumd
3. Spontaeous PROM as confirmed by history and sterile speculum examination
4. modified bishop score <6
5. no detectable uterine contractions on admission
6. clear liqour and duration of PROM <6 hours at admission

Exclusion Criteria:

1. meconium stained liqour
2. patients with features of chorioamnionitis (fever , tachycardia, abdominal tendernessor foul smeeling vaginal discharge
3. maternal medical diseaseincluding prompt delivery or C section like severe preeeclampsia, renal or cardiac disease
4. presence of contraindications to labour such as placenta previa , Vasa previa,previous uterine surgery (e.g myomectomy ) that increases the risk of uterine rupture , previous C section
5. history of antepartum hemorrhage
6. Moderate to severe IUGR as diagnosed on ultrasound and doppler studies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 88 (Actual)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Duration of labour | 24 hours
  the duration of labour was assesed after each method of induction when patients presented with PROM

SECONDARY OUTCOMES:
Frequency of Normal Vaginal Delivery | 24 hours
  Frequency of having a vaginal delivery was calculated in each interventional group

CONTACTS AND LOCATIONS:
Locations (1):
- Hameed Lateef Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The participants have not given the cosent to share their personal data